CLINICAL TRIAL: NCT00831142
Title: Characterization of Prostate Cancer With 3T MR
Status: Active, not recruiting | Type: Observational
Sponsor: Beth Israel Deaconess Medical Center (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, David Alsop, Director of MR Research, Beth Israel Deaconess Medical Center
Other Study IDs: 2006P000154; 5R01CA116465-04 (NIH)
Record Dates: First submitted 2009-01-27; First posted 2009-01-28 (Estimated); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; MRI; Prostatectomy
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Prostate Cancer: Males with prostate cancer, referred for biopsy or radical prostatectomy

SUMMARY:
The long-term goal of this proposal is to provide a pre-treatment evaluation that can assist in the rational selection of patients to undergo appropriate and definitive therapy for prostate cancer. In so doing, it may be possible to further improve the numbers and percentage of cancer patients who receive effective therapy that will cure the disease and maximize their quality of life following therapy.

* Aim 1: To evaluate the accuracy of T2W MRI, DCE-MRI and their combined data for staging prostate cancer.
* Aim 2: To evaluate the accuracy of MRI in determining tumor volume in the prostate gland.
* Aim 3: To evaluate the accuracy of MRI in grading prostate cancer.

DETAILED DESCRIPTION:
In our laboratory we have combined the use of new 3T clinical magnetic resonance (MR) technology, dynamic-contrast enhancement (DCE), and a unique endorectal-coil (ERC) probe in order to non-invasively obtain images of the prostate gland with higher signal-to-noise resolution and better spectral dispersion than has been previously achieved. This imaging strategy acquires higher-resolution images with smaller voxel sizes than has been possible with prior MR technology and more comprehensive tissue sampling compared to other pre-surgical assessments. This methodology should make it feasible to assess prostate-tissue morphology and additional features of prostate cancer such as tissue metabolism, tissue kinetics, and the vascular microenvironment, and thus provide a non-invasive tool to: 1) detect extra-capsular spread, 2) detect specific areas within the prostate that harbor cancer, 3) determine the aggressiveness of the cancer and 4) direct biopsy and treatment specifically to diseased areas.

In order to prospectively validate these goals we will recruit successive patients who have been scheduled for prostate removal to participate to our protocol. Each patient will be studied with an ERC MRI at 3T using T2-weighted (T2W) imaging, DCE 3D T1-weighted imaging and MR spectroscopy (MRS). A pathologist using whole mount preparations will independently analyze each patient's prostate specimen. The whole mount data will be used as the standard against which we will compare the observations and data obtained from the 3T MRI findings.

Aim 1: To evaluate the accuracy of T2W MRI, DCE-MRI and their combined data for staging prostate cancer.

Supplementing T2W imaging with the high-resolution capability of 3TMR, we will apply standard morphologic criteria used at 1.5T to determine the presence or absence of extracapsular extension (ECE) of disease. The possible incremental value of high spatial resolution, dynamic contrast-enhanced data will be investigated. MRI results will be compared to ECE determination at whole-mount pathology.

Aim 2: To evaluate the accuracy of MRI in determining tumor volume in the prostate gland.

Using dynamic-contrast enhanced MRI with parametric analyses and T2-weighted images, both at smaller voxel sizes than have been used previously, will be our approach. Tumor volumes determined with MRI will be compared to those determined at pathology.

Aim 3: To evaluate the accuracy of MRI in grading prostate cancer.

The enhanced resolution available at 3T offers new opportunities to compare Gleason grades with independent and combined assessments of tissue kinetics and metabolism. Pixel by pixel parametric analyses will be obtained. Furthermore, choline to citrate and choline plus creatine to citrate ratios determined using MRS techniques will be obtained. Single voxel techniques will first be employed, followed by 3D chemical shift imaging, when the latter becomes available at 3T. DCE and MRS data will be compared both separately and in combination to the histologic Gleason scores of the comparable tumor identified at whole mount pathology.

ELIGIBILITY:
Inclusion Criteria

1. Biopsy-proven adenocarcinoma of the prostate.
2. Written documentation from the urologist stating the anticipation that the patient will undergo radical prostatectomy or biopsy of the prostate within six months of MRI.
3. The interval between biopsy and protocol MRI must not be less than 2 weeks.
4. Pathologic specimens from radical prostatectomy must be provided for whole mount analysis.
5. Patients will sign a study-specific consent prior to study entry.
6. Men above the age of 40 years old

Exclusion Criteria

1. Patients who because of age, general medical or psychiatric condition, or physiologic status unrelated to the presence of prostate cancer cannot give valid informed consent.
2. Patients unwilling or unable to undergo MRI including patients with contra-indications to MRI such as the presence of cardiac pacemakers or non-compatible intracranial vascular clips.
3. Patients who cannot tolerate or have contra-indications to ERC insertion; for example, patients who have had a prior abdominoperineal resection of the rectum or have Crohn's disease.
4. Patients with an allergic reaction to latex.
5. Cryosurgery, surgery for prostate cancer including TURP, prostatic radiotherapy, including bradiotherapy for rectal cancer, androgen deprivation therapy, rectal surgery, or alternative medicine prior to radical prostatectomy.
6. Any metallic implant (e.g. hip) or device that might distort local magnetic field and compromise quality of MRI.
7. Radical prostatectomy or biopsy of the prostate not planned to be performed within six (6) months of protocol MRI.
8. Patients who have undergone BCG for bladder cancer.
9. Patients with severe motion artifacts rendering the data unusable.
10. Patients who have an allergic history to gadopentetate dimeglumine administration.
11. Patients with a contraindication to the administration of glucagon (pheochromocytoma, islet pancreatic tumor, or insulin-dependent diabetes) or a prior history of allergic reaction following glucagon administration.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The sample will include 50 male patients per year of all races and ethnic origins over 40 years of age who are likely to undergo radical prostatectomy for prostate carcinoma. Patients will be imaged using MRI/MRS.
Sampling Method: Non-Probability Sample
Enrollment: 236 (Actual)
Dates: Start 2006-06; Primary Completion 2012-01 (Actual); Study Completion 2025-05-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: David C Alsop, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States